CLINICAL TRIAL: NCT06938529
Title: A Phase I Pharmacokinetic Study of VCT220 in Subjects With Varying Degrees of Hepatic Impairment and Normal Hepatic Function
Brief Title: A Pharmacokinetic Study of VCT220 in Particicants With Hepatic Injury and Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vincentage Pharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VCT220-I-05
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Obesity, Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Subjects with mild hepatic impairment (Child-Pugh Class A, score of 5-6)
  Interventions: Drug: VCT220
- Group B (Experimental): Subjects with moderate hepatic impairment (Child-Pugh Class B, score of 7-9)
  Interventions: Drug: VCT220
- Group C (Placebo Comparator): Subjects with normal hepatic function matched to hepatic impairment subjects
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VCT220 — Small molecule GLP-1RA tablet, film coated
  Arms: Group A; Group B
Drug: Placebo — VCT220 Placebo tablet
  Arms: Group C

SUMMARY:
This is an open-label, non-randomized study to assess how VCT220 is absorbed, distributed, metabolized, and eliminated after a single oral dose. The study includes three groups: subjects with mild hepatic impairment (Child-Pugh Class A), subjects with moderate hepatic impairment (Child-Pugh Class B), and healthy subjects matched by gender, age, and body mass index (BMI). It will also explore the relationship between baseline liver function measures and the pharmacokinetic (PK) parameters of VCT220, to support appropriate dosing recommendations for patients with liver impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must fully understand the purpose and requirements of the study, voluntarily participate in the clinical trial, sign a written informed consent form, and be able to complete the entire study process as required;
2. Subjects must be between 18 and 75 years old (inclusive), of any sex;
3. At screening, male subjects must weigh ≥50 kg and female subjects must weigh ≥45 kg, with a body mass index (BMI = weight (kg)/height² (m²)) between 18.5 and 35.0 kg/m² (inclusive);
4. Subjects and their partners must agree to have no plans for pregnancy or sperm/egg donation from the signing of the informed consent form until 6 months after the last administration of the study drug, and must voluntarily use effective contraception.

For subjects with hepatic impairment, the following additional inclusion criteria must be met:

1. Subjects must have hepatic impairment caused by a primary liver disease, classified as Child-Pugh Class A (score 5-6) or Class B (score 7-9) at screening, and must not have used albumin within 14 days prior to screening. The hepatic impairment must be confirmed as stable (≥1 month) based on medical history, physical examination, laboratory tests, or imaging studies;
2. Subjects must not have taken any medications within 1 week prior to screening, or, if long-term treatment for hepatic impairment and/or other comorbidities is necessary, must have been on a stable regimen for at least 4 weeks prior to screening (stable medication use to be determined by the investigator, excluding prohibited medications per protocol).

Exclusion Criteria:

* Known allergy to any component of the investigational drug, similar drugs (GLP-1 receptor agonists), or their excipients, a history of allergic constitution (multiple drug and food allergies), or a history of allergic diseases (such as asthma, urticaria, eczema, etc.);
* A history of hypoglycemia;
* Personal or family history of medullary thyroid carcinoma (MTC) or type 2 multiple endocrine neoplasia syndrome (MEN2), or suspected MTC as judged by the investigator;
* A history of pancreatitis (chronic or acute pancreatitis);
* A history of malignant tumors or malignancy within the past 5 years (excluding stable liver cancer post-surgery for ≥2 years, treated and non-recurrent skin non-melanoma cancers, and removed cervical intraepithelial neoplasia);
* Severe infection, trauma, gastrointestinal surgery, or other major surgeries within the 4 weeks prior to screening;
* Clinically significant abnormalities on a 12-lead electrocardiogram (ECG), such as tachycardia/bradycardia requiring medication, second to third-degree atrioventricular block, QTcF interval prolongation (QTcF >470 ms in males, >480 ms in females) as per Fridericia's formula, or other clinically significant abnormalities as determined by the clinician;
* Estimated glomerular filtration rate (eGFR) <60 ml/min/1.73m², calculated using the Modification of Diet in Renal Disease (MDRD) formula;
* Hemoglobin A1c (HbA1c) >6.5% at screening;
* Plans to undergo surgical treatment during the trial or a tendency to require hospitalization;
* Positive HIV antibody (HIV-Ab) test.
* Used enzyme inducers or inhibitors (strong and moderate inducers and inhibitors of CYP3A4, strong inducers and inhibitors of CYP2C8 and CYP2D6) within 4 weeks prior to dosing;
* Took any medication (including traditional Chinese medicine, vitamins, supplements) within 14 days prior to dosing (or 5 half-lives, whichever is longer), except for stable medication use in subjects with hepatic impairment;
* Participated in another clinical trial and received investigational drugs or medical devices within 1 month prior to screening, with the last dose date of the clinical study as the baseline (if the clinical trial drug has a long half-life, there should be at least a 5 half-life gap between this study and the previous one);
* Lost blood or donated ≥400 mL of blood within 3 months prior to dosing, or plans to donate blood within 1 month after the trial ends;
* A smoker or has smoked more than 5 cigarettes daily in the 3 months prior to screening, or unable to stop tobacco product use during the study;
* Currently or frequently consumes alcohol, i.e., females drinking more than 7 units of alcohol per week, males drinking more than 14 units of alcohol per week (1 unit = 285 mL beer, 25 mL of 40% alcohol, or 100 mL of wine); or testing positive for alcohol on a breathalyzer test at baseline, or unable to abstain from alcohol during the study;
* Abused drugs or used soft drugs (e.g., cannabis) within 3 months prior to dosing, or used hard drugs (e.g., cocaine, amphetamines, piperazines) within 1 year prior to dosing, or tested positive for drug abuse on baseline urine screening;
* Consumed grapefruit juice/grapefruit, methylxanthine-containing foods or drinks (tea, coffee, cola, chocolate, energy drinks), or other substances affecting drug absorption, distribution, metabolism, or excretion within 48 hours prior to dosing;
* Unable to tolerate venipuncture or experiences fainting or anxiety with needles or blood;
* Received a vaccination within 1 month prior to screening;
* Pregnant or breastfeeding women, or tested positive for a blood pregnancy test;
* The investigator considers the subject to have poor compliance, or other factors that make them unsuitable for participation in the study.

Additional exclusion criteria for subjects with liver dysfunction (exclude if any one condition is met):

1. Positive syphilis test result;
2. History of liver transplantation;
3. Drug-induced liver injury;
4. Acute liver injury caused by various reasons;
5. Cholestatic liver disease;
6. Liver failure with any of the following conditions: Uncontrollable infection; Grade 3/4 hepatic encephalopathy;
7. Severe complications of cirrhosis with any of the following conditions: Active bleeding from esophageal or gastric varices; Severe/late-stage ascites or pleural effusion requiring puncture, drainage, and albumin supplementation; Hepatorenal syndrome subjects, or those deemed unsuitable for participation in the study by the investigator;
8. Poorly controlled hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg), heart rate >120 bpm (allowing for two re-tests);
9. History of any serious illness other than the primary liver disease itself, or a history or clinical laboratory abnormalities (including but not limited to circulatory, endocrine, neurological, digestive, urinary, hematologic, immune, psychiatric, and metabolic diseases) that may affect the study results, as determined by the investigator;
10. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) levels >5 times the upper limit of normal (ULN) during the screening period.

Additional exclusion criteria for subjects with normal liver function (exclude if any one condition is met):

1. Positive test result for Treponema pallidum (TP) antibody;
2. History of significant primary organ disease, including but not limited to neurological, psychiatric, cardiovascular, gastrointestinal, respiratory, urinary, endocrine, hematological, or immune diseases, as judged by the investigator to be unsuitable for participation in this trial;
3. History of liver dysfunction or abnormal screening results (including physical examination, vital signs, blood routine, urine routine, blood biochemistry, coagulation function, 12-lead ECG, chest X-ray, abdominal ultrasound, etc.) deemed clinically significant by the investigator;
4. Age outside of the mean ±10 years for subjects with mild/moderate liver dysfunction, and/or BMI outside of the ±10% of the mean BMI for subjects with mild/moderate liver dysfunction;
5. Positive for hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody during the screening period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-04-18 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of VCT220 | Predose up to 72 hours postdose (D1 to D4)
Area Under the Serum Concentration Curve From Time 0 to the Last Measurable Concentration (AUC0-last) of VCT220 | Predose up to 72 hours postdose (D1 to D4)
Area Under the Serum Concentration Curve From Time 0 to Infinity(AUC0-inf) of VCT220 | Predose up to 72 hours postdose (D1 to D4)

SECONDARY OUTCOMES:
Safety evaluation endpoints | From Day 1 to Day 10
  Including the incidence and severity of AEs and SAEs.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No